CLINICAL TRIAL: NCT00779285
Title: Cardiac Safety Profile of Caelyx Therapy in Anthracyclin Pretreated Metastatic Breast Cancer Patients.
Brief Title: Safety Study of CAELYX in Patients With Metastatic Breast Cancer Previously Treated With Anthracyclines (Study P04057)(TERMINATED)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P04057; EUDRACT NO. 2004-001177-25
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Results first posted 2010-03-10 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-06

CONDITIONS: Breast Neoplasm
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-arm (Experimental): Pegylated Lyposomal Doxorubicin (Caelyx) 50 mg/m2, given for 6 cycles
  Interventions: Drug: Pegylated Liposomal Doxorubicin

INTERVENTIONS:
Drug: Pegylated Liposomal Doxorubicin — Pegylated Liposomal Doxorubicin (Caelyx) IV, 50 mg/m2 once every 4 weeks for 6 cycles or until disease progression, whichever is earlier. Patients still receiving clinical benefit after a total of 6 cycles of Caelyx, may continue therapy at the discretion of the investigator.
  Other Names: SCH 200746

SUMMARY:
The purpose of this study is to evaluate the cardiac safety of Caelyx in patients with metastatic breast cancer who have previously received chemotherapy with anthracyclines.

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically or cytologically confirmed metastatic breast cancer (no prior chemotherapy for metastatic disease).
* Prior treatment with an anthracyclin-containing regimen in the adjuvant setting (cumulative dose >240mg/m^2 and <360mg/m^2 doxorubicin or >430mg/m^2 and <650mg/m^2 epirubicin).
* Women >18 years of age.
* Documented measurable and/or evaluable metastatic breast cancer by appropriate radiological imaging (computed tomography (CT) scan and/or magnetic resonance imaging (MRI)).
* Performance status of at least 60% (Karnofsky index) and a life expectancy of at least 12 weeks.
* Left ventricular ejection fraction >50%.
* Normal organ function, except if abnormal due to tumor involvement.

  * Adequate bone marrow function as indicated:

    * Platelets >100,000/mm^3
    * Hemoglobin >9 g/dL
    * Neutrophils >1,500/mm^3
  * Adequate renal function as indicated by:

    * Serum Creatinine <1.5 x the upper limit of normal
  * Adequate liver function, as indicated by:

    * Bilirubin and aspartate aminotransferase (AST) or alanine aminotransferase (ALT) <2 times upper limit of normal (<4 times upper limit of normal when related to primary disease)
* Subjects must be capable to demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent.
* Women of childbearing potential (includes women who are less than 1 year postmenopausal and women who become sexually active) must be using an acceptable method of birth control (e.g., hormonal contraceptive, medically prescribed intrauterine device (IUD), condom in combination with spermicide) or be surgically sterilized (e.g., hysterectomy or tubal ligation).
* Subjects must understand and be able to adhere to the dosing and visit schedules.

Exclusion Criteria:

* Patient is pregnant or is breastfeeding.
* Patients with moderate or severe heart failure (New York Heart Association (NYHA) class III/IV).
* Hypersensitivity to anthracycline therapy or a history of severe hypersensitivity reactions to products containing Cremophor® EL (e.g., cyclosporin for injection concentrate and teniposide for injection concentrate).
* Prior chemotherapy for metastatic disease.
* Clinically significant hepatic disease (except liver metastases of primary disease).
* Uncontrolled bacterial, viral, or fungal infection.
* Radiotherapy in the last 4 weeks or prior radiation therapy to more than one-third of the hemopoietic sites.
* Any other currently known malignancy or pre-malignant lesions or any history of other malignancy within the past five years (except non-melanoma skin cancer and surgically cured cervical cancer).
* Symptomatic brain metastasis.
* Patients who are incapacitated, largely or wholly bedridden or confined to a wheelchair, and who have little or no ability for self-care.
* Current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, endocrine, pulmonary, cardiac, neurological or cerebral disease.
* Documented human immunodeficiency virus (HIV) infection.
* Any condition (medical, social, psychological) which would prevent adequate follow-up.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2006-02; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Caelyx: Pegylated Lyposomal Doxorubicin (Caelyx) 50 mg/m2, given for 6 cycles
Period: Overall Study
Arm/Group | Caelyx
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Caelyx
Number analyzed (Participants) | 1
Age, Customized [Number; unit: participants] | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  Hungary | 1

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Events
Description: A cardiac event was defined as a decrease in left ventricular ejection fraction (LVEF) of >=20 points from baseline if the resting LVEF remained in the normal range, or a decrease of >=10 points if the LVEF became abnormal (lower than the institutional lower limit of normal).
Time Frame: Every 4 weeks during 6 cycles.
Measure: Number; unit: Cardiac Events
Arm/Group | Caelyx
Number analyzed (Participants) | 1
Cardiac Events | 0

ADVERSE EVENTS:
Arm/Group | Caelyx
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caelyx (N=1)
Maculopapulosus exanthema (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigator agrees not to publish/publicly present any

interim results without prior Sponsor written consent and agrees to provide 30 days written notice prior to submission to permit review of abstracts/manuscripts which report any results. Sponsor has the right to review/comment/edit to ensure confidentiality, information accuracy, and that the presentation is fairly balanced. If the parties disagree, the investigator agrees to meet with Sponsor to discuss/resolve any disagreement.